CLINICAL TRIAL: NCT05401214
Title: Pre-Approval Access Single Patient Request for Niraparib / Abiraterone Acetate Combination (Nira/AA Combination)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR109197; 67652000MPC4002 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-05-27; First posted 2022-06-02 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Castration-resistant Prostate Cancer
MeSH Terms: interventions — niraparib; Abiraterone Acetate; Prednisone; Prednisolone

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Niraparib plus Abiraterone Acetate (Nira/AA) combination — Nira 100 milligrams (mg)/AA 500 mg combination will be administered orally as immediate-release film coated tablets.
Drug: Prednisone/Prednisolone — Prednisone/Prednisolone 10 mg will be administered orally.

SUMMARY:
The purpose of this pre-approval access is to provide Niraparib plus Abiraterone Acetate (Nira/AA combination) in the treatment of (a) participant(s) with first line metastatic castration-resistant prostate cancer with specific Homologous Recombination Repair (HRR) gene alterations.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with metastatic castration-resistant prostate cancer (mCRPC)
* A confirmed homologous recombination repair (HRR) gene alteration as identified by a genomic assay through use of a validated test
* Eastern Cooperative Oncology Group Performance Score (ECOG PS) Grade of 0 or 1
* Willing to receive concomitant prednisone/ prednisolone 10 milligrams (mg) (not provided by Janssen) daily while receiving niraparib/abiraterone acetate (Nira/AA) combination treatment
* Willing to continue treatment with gonadotropin-releasing hormone (GnRH) analogue if not surgically castrated

Exclusion Criteria:

* Prior treatment with a Poly ADP-ribose Polymerase (PARP) inhibitor
* Prior systemic therapy for mCRPC (that is, taxane-based chemotherapy, androgen signaling inhibitors). Ongoing androgen deprivation therapy (ADT), prior systemic treatment (example, apalutamide, enzalutamide, darolutamide, docetaxel) for earlier disease settings (example, hormone sensitive disease, non-metastatic castration-resistant disease); and treatment recently initiated with abiraterone acetate for mCRPC less than or equal to (<=) 60 days is permitted
* Other treatment options available or participant eligible or able to participate in a clinical trial for first line mCRPC with HRR gene alterations
* Moderate-severe pain
* History or current diagnosis of myelodysplastic syndrome (MDS)/acute myeloid leukemia (AML)

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC